CLINICAL TRIAL: NCT01164436
Title: French Cohort of HIV Associated Lymphomas
Brief Title: Cohort of HIV Associated Lymphomas
Acronym: ANRS CO16
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Dr Yassine Taoufik Dr Houria Chavez Hôpital Bicêtre CIB Paris Sud France (Unknown); Dr Guislaine Garcelain Hôpital Pitié Slapétrière Paris France (Unknown); University Hospital, Grenoble (Other); Dr Irène Joab Hôpital Paul Brousse Villejuif France (Unknown); Dr Alex Duval Fondation Jean Dausset CEPH (Unknown); Hopital Antoine Beclere (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-AO0258-45
Record Dates: First submitted 2009-12-22; First posted 2010-07-16 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The incidence of lymphomas is increased among HIV infected patients. In 70 % of cases, those are Non Hodgkin's lymphomas (NHL) and Hodgkin lymphomas (HL) in 30% of cases. In France, their incidence is estimated to 100 cases per year (data from the "Base de données Hospitalière Française sur l'Infection à VIH" (FHDH)). The main mechanisms involved in lymphomagenesis are immune dysfunction, involvement of oncogenic viruses (Epstein-Barr (EBV) and HHV8) and molecular oncogenic events. A better understanding of these different pathways, give the possibility to design specific treatments. The treatment of these lymphomas is not standardized. A prospective study of patients with HIV associated lymphoid malignancies is an innovating tool to answer epidemiological, physiopathological and therapeutic questions. We propose a prospective multicentric study of these patients.

The main objectives of this prospective study are to:

* evaluate the incidence, characterise clinically and histologically NHL and HL cases associated to HIV
* perform an observational study of the treatment and outcome of these patients out of the context of clinical trials,
* study the differentiation and activation of B-cell populations,
* better understand the role of specific T cell responses in the control of EBV infection,
* allow other biological studies from the ANRS group " Lymphome et VIH ".

The recruitment of 40 cases per year is expected. The length of inclusions is 7 years. The follow-up will be of 2 years. Clinical, pathological and biological data at diagnosis and during follow-up will be collected. This will allow characterizing the lymphoma, the HIV infection, the antitumoral treatments and the outcome of lymphoma. Biological samples will be centralized to collect cell, DNA, RNA, plasma, serum and tumour collections (Y.Taoufik, S Prevot* ). To better understand the EBV infection and lymphomagenesis in HIV infection, we propose to follow the viral load and the molecular characteristics of EBV in PBMC, plasma and tumour (P.Morand* , V.Boyer* ), to investigate the EBV-T cell responses (G.Carcelain) and the presence and reactivation of EBV in peripheral B cells (C.Amiel* , JC Nicolas) and in tumoral samples (M.Raphael* , I.Joab* ). The other mechanisms of lymphomagenesis in HIV infection will be studied by the analysis of the sub-populations of B-cells in terms of activation and differentiation (Y.Taoufik) and by the characterization of MSI tumours (A.Duval).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients over 18 years of age
* patients with HIV-1 or 2 infection
* with Non Hodgkin's lymphomas (NHL) or Hodgkin lymphomas (HL) in the diagnosis or in relapse
* sign an informed consent

Exclusion Criteria:

* patients who suffered from acute leukemia
* patients treated for lymphoïd blood disease
* Patients whose lymphomas treatment was stopped for less than 3 months
* unaffiliated to the social healthy security french system

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The recruitment of 80 cases per year is expected. The length of inclusions is 5 years. The follow-up will be of 5 years. Clinical, pathological and biological data at diagnosis and during follow-up will be collected. This will allow characterizing the lymphoma, the HIV infection, the antitumoral treatments and the outcome of lymphoma. Biological samples will be centralized to collect cell, DNA, RNA, plasma, serum and tumour collection.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2008-06; Primary Completion 2015-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Correlation between EBV viral load and plasma HIV RNA viral load and CD4 cell count in HIV-infected patients with lymphomas (LNH or LH) at the time of lymphoma diagnosis | 5 year

SECONDARY OUTCOMES:
Survival rate in HIV patients with NHL or HL | 5 year
Progression-free survival rate in HIV patients with NHL or HL | 5 year
Levels of EBV in tumors of HIV patients with NHL or HL | 5 year
  measurement of EBV using in situ hybridization applied to paraffin sections
Levels of B cell activating cytokines in plasma of HIV patients with NHL or HL | 5 year
  measurement of concentrations of IL-6, IL-10, BAFF in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Caroline BESSON, Principal Investigator — Service Hématologie Immunologie Biologie, Hopital Bicetre; Gilles Pialoux, PH, Principal Investigator — Hôpital Tenon Paris; Marie Caroline Meyonas, PH, Principal Investigator — Hôpital St Antoine Paris; Christine Katlama, PH, Principal Investigator — Hôpital Pitiè Salpétrière; Jean Gabarre, MD, Principal Investigator — Hôpital Pitiè Salpétrière Paris; Dominique Salmon, PH, Principal Investigator — Hôpital Cochin PARIS; François Dreyfus, PH, Principal Investigator — Hôpital Cochin Paris; Jean Paul Viard, PH, Principal Investigator — Hotel Dieu PARIS; Alain Devidas, PH, Principal Investigator — Corbeil Essone 91; Emma Goldschmidt, MD, Principal Investigator — Villejuif 94; Cecile Goujard, MD, Principal Investigator — Hôpital Bicêtre 94; Laurent Blum, MD, Principal Investigator — Pointoise 95; François Boué, PH, Principal Investigator — Clamart 92; Eric Rosenthal, MD, Principal Investigator — Nice 06; Christine Burty, MD, Principal Investigator — Vandoeuvre les Nancy 54; Jean Marie Lang, PH, Principal Investigator — Strasbourg 67; Renaud Verdon, PH, Principal Investigator — Caen 14; Yazdan Yazdanpanah, PH, Principal Investigator — Tourcoing 59; Christine Drobacheff, MD, Principal Investigator — Besancon 25; Bruno Marchou, PH, Principal Investigator — Toulouse 31; Corinne Couteau, MD, Principal Investigator — Toulouse 31; Philippe Morlat, PH, Principal Investigator — Bordeaux 33; Christian Trepo, PH, Principal Investigator — Lyon 69; Hervé Ghesquières, PH, Principal Investigator — Lyon 69; Régis Costellos, PH, Principal Investigator — Marseille; Bertrand Coiffier, Ph, Principal Investigator — Pierre Bénite; Claude Beuscart, MD, Principal Investigator — St Brieuc 22; Philippe Perre, MD, Principal Investigator — La Roche Sur Yon 85; Patrice Poubeau, MD, Principal Investigator — St Pierre 97; François Raffi, PH, Principal Investigator — Nantes 44; Frédéric Lucht, PH, Principal Investigator — St Etienne 42; Nicolas Mounier, PH, Principal Investigator — Nice 06; Cédric Arvieux, PH, Principal Investigator — Rennes 35; Serge Herson, PH, Principal Investigator — Pitié Salpétrière Paris; Jean François Bergmann, PH, Principal Investigator — Lariboisière Paris; André Cabié, PH, Principal Investigator — Fort de France 97( Martinique)
Locations (1):
- BESSON, Paris, France

REFERENCES:
- [Derived] Lievin R, Maillard A, Hendel-Chavez H, Krzysiek R, Lancar R, Algarte-Genin M, Costagliola D, Assoumou L, Taoufik Y, Besson C. Immune reconstitution and evolution of B-cell-stimulating cytokines after R-CHOP therapy for HIV-associated DLBCL. Blood Adv. 2024 Dec 10;8(23):6017-6027. doi: 10.1182/bloodadvances.2024014116. PMID 39348664